CLINICAL TRIAL: NCT00954096
Title: The Effect Of Nicotine On Indices Of Arterial Function And Oxidative Stress
Brief Title: Nicotine Patch, Blood Flow and Oxidative Stress Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Garret A. FitzGerald M.D Chair, Department of Pharmacology- Director, Institute for Translational Medicine and Therapeutics, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 707275; 0875
Record Dates: First submitted 2009-07-29; First posted 2009-08-06 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal nicotine patch or placebo (Experimental): A single blood specimen (85ml) will be drawn. They will be asked to empty their bladder. The patch will be applied. Following application of the patch, heart rate and blood pressure will be measured every 15 minutes for the 1st hour, every 30 minutes for the next 3 hours and hourly after that until the end of the study. Urine will be collected in two 4-hour aliquots. FMD will be measured after approximately 6 hours of nicotine exposure. After 8 hours exposure, following the end of the 2nd urine collection, the patch will be removed and the subject discharged. Following a minimum of 2 weeks (maximum 8 weeks) washout, the subject will repeat the study, receiving the other patch.
  Interventions: Drug: transdermal nicotine patch (7mg)

INTERVENTIONS:
Drug: transdermal nicotine patch (7mg) — A 7mg transdermal nicotine patch will be applied to the subject's arm for an 8 hour period.
  Other Names: Nicotine patch; Habitrol; Nicoderm CQ; Nicotrol

SUMMARY:
This study will address the hypothesis that nicotine, like cigarette smoking acting as a pro-oxidant may have adverse effects on arterial function.

DETAILED DESCRIPTION:
Smoking causes >400,000 deaths from cardiovascular disease (CVD) per year. The molecular basis of smoking induced tissue injury remains unclear but considerable evidence supports a role for oxidant stress (OS).

Arterial function has been shown to be impaired in smokers even before the onset of angiographically demonstrable atherosclerosis. Defects in endothelium dependant flow mediated vasodilatation (FMD) are seen in those at risk of or with overt vascular disease.

Cigarette smoking is highly addictive. Spontaneous quit rates approximate 3%. Even those using nicotine replacement therapy (NRT) have high relapse rates (67-75%) on completion of the 8-12 week course of NRT. Thus there is interest in the use of extended NRT as a "safer" alternative to cigarette smoking. However such assumptions may be premature. Nicotine demonstrates proxidant effects in vitro and in small studies has been associated with endothelial dysfunction. Studies simultaneously assessing the effects of nicotine on oxidative stress and arterial function in humans have not been performed.

The current proposal will address the hypothesis that nicotine, like cigarette smoking acting as a pro-oxidant may have adverse effects on arterial function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Nonsmokers who have never smoked
* Normal medical history
* Normal physical examination
* Normal laboratory data
* Negative urinary pregnancy test for females

Exclusion Criteria:

* Previous CVD
* Chronic medication use
* History alcoholism
* History of smoking
* Current pregnancy
* Subjects, who have less than or equal to 60% platelet aggregation in response to arachidonic acid will also be excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2002-10; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Assess the dose-related effects of nicotine in humans, on novel indices of lipid peroxidation, protein oxidation and DNA modification by lipid adducts. | 1 - 3 years

SECONDARY OUTCOMES:
Assess the dose-related effects of nicotine in humans on COX activation. | 1 year
Assess the dose-related effects of nicotine in humans on blood flow mediated arterial function. | 3 - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania Institute for Translational Medicine and Therapeutics
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Institute for Translational Medicine and Therapeutics, University of Pennsylvania — http://www.itmat.upenn.edu/